CLINICAL TRIAL: NCT06238622
Title: An Open-label Extension Trial of the Long-term Safety and Efficacy of BI 1015550 Taken Orally in Patients With Idiopathic Pulmonary Fibrosis (IPF) and Progressive Pulmonary Fibrosis (PPF) (FIBRONEER™-ON)
Brief Title: A Follow-up Study to Test Long-term Treatment With Nerandomilast in People With Pulmonary Fibrosis Who Took Part in a Previous Study With Nerandomilast
Acronym: FIBRONEER™-ON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0031; 2023-507353-15-00 (Other: CTIS)
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis; Progressive Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BI 1015550 treatment group (Experimental)
  Interventions: Drug: Nerandomilast

INTERVENTIONS:
Drug: Nerandomilast — Nerandomilast
  Other Names: BI 1015550, JASCAYD®

SUMMARY:
This study is open to people with idiopathic pulmonary fibrosis (IPF) or progressive pulmonary fibrosis (PPF). They can only take part if they have completed treatment in a previous study with a medicine called nerandomilast or BI 1015550.

The goal of this study is to find out how well people with pulmonary fibrosis tolerate long- term treatment with nerandomilast. The study also tests whether nerandomilast improves lung function and prolongs the time until symptoms get worse, participants need to go to the hospital, or die.

Every participant takes nerandomilast as tablets for up to 1 year and 10 months. The participants may also continue their regular treatment for pulmonary fibrosis during the study.

Participants visit their doctors regularly. During these visits, the doctors collect information on any health problems of the participants. Participants also regularly do lung function tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed treatment in the parent trials (1305-0014, 1305-0023, or 1305-0035) without prematurely discontinuing treatment permanently according to protocol (i.e. completed treatment with or without temporary treatment interruption)
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
3. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. WOCBP taking oral contraceptives (OCs) also have to ensure the use of one barrier method during sexual intercourse with their partner, e.g., condom to account for the risk of potentially reduced efficacy of the OCs in the event of severe vomiting and diarrhoea. For France, fertile males must be ready and able to use acceptable methods of birth control

Exclusion Criteria:

1. Any disease that may put the patient at risk when participating in this trial at investigator's discretion.
2. Patient exhibits suicidality, in the clinical judgment of the investigator or according to the following criteria at Visit 1:

   * any suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
   * any suicidal ideation of type 4 or 5 in the Columbia-Suicide Severity Rating Scale (C-SSRS) (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)
3. Patients with clinically relevant severe depression at investigator's discretion or a Hospital Anxiety and Depression Scale (HADS) subscore >14 at Visit 1.
4. An occurrence of malignant neoplasm other than appropriately treated basal cell carcinoma or in situ squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix at Visit 1.
5. Patient will undergo lung transplantation, with an assigned date of surgery.
6. Patients with a Body Mass index (BMI) <18.5 kg/m² that experienced an additional, unexplained and clinically significant (>10%) weight loss during the parent trial
7. At Visit 1, patients with ongoing Adverse Event of Special Interest (AESI), except for latent tuberculosis (suspected vasculitis, Drug Induced Liver Injury (DILI), severe infections) that led to temporary treatment interruption in the parent trial
8. Patients who must or wish to take restricted medications or any drug considered likely to interfere with the safe conduct of the trial.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any adverse event over the course of the extension trial (yes/no) i.e. up until the follow-up/end of study visit planned at the latest at week 99 | Up to 99 weeks and 3 days

SECONDARY OUTCOMES:
Absolute change from baseline in Forced vital capacity (FVC) (mL) over time | Up to 98 weeks
Absolute change from baseline in % predicted in Forced vital capacity (FVC) over time | Up to 98 weeks
Time to absolute decline in FVC % predicted of >10% from baseline over the duration of the trial | Up to 98 weeks
Time to first acute Idiopathic Pulmonary Fibrosis/Progressive Pulmonary Fibrosis (IPF/PPF) exacerbation, first hospitalisation for respiratory cause, or death (whichever occurs first) over the duration of the trial | Up to 98 weeks
Time to first acute Idiopathic Pulmonary Fibrosis/Progressive Pulmonary Fibrosis (IPF/PPF) exacerbation or death over the duration of the trial | Up to 98 weeks
Time to hospitalisation for respiratory cause or death over the duration of the trial | Up to 98 weeks
Time to absolute decline in Forced vital capacity (FVC) % predicted of >10% from baseline or death over the duration of the trial | Up to 98 weeks
Time to relative decline in Forced vital capacity (FVC) % predicted of >10% from baseline or death over the duration of the trial | Up to 98 weeks

CONTACTS AND LOCATIONS:
Locations (372):
- United States (57):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Clinical Research Specialists LLC - Kissimmee, Kissimmee, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Piedmont Physicians Pulmonary & Sleep Medicine of Buckhead, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Northshore University Health System, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Creighton University, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Northern Westchester Hospital, Mount Kisco, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Research Center-Winston Salem-69289, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Infinity Medical Research, Inc., East Providence, Rhode Island
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Clinical Trials Center of Middle Tennessee, LLC, Franklin, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Intermountain Medical Center-Murray-69497, Murray, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (9):
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Consultorios Médicos del Buen Ayre, Capital Federal
  - CEMER-Centro Medico De Enfermedades Respiratorias, Florida
  - Instituto Ave Pulmo, Mar del Plata
  - INSARES, Mendoza
  - Centro Respiratorio de Quilmes, Quilmes
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
- Australia (11):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Lung Research Queensland, Chermside, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Trialswest, Spearwood, Western Australia
  - Macquarie University, Macquarie Park
- Austria (5):
  - Krems University Hospital, Krems
  - LKH Salzburg University Hospital, Salzburg
  - AKH - Medical University of Vienna, Vienna
  - Clinic Floridsdorf, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (7):
  - Ziekenhuis Netwerk Antwerpen (ZNA) - Campus Middelheim, Antwerp
  - ULB Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Brazil (9):
  - Serviços Medicos Respirar Sul Fluminense, Barra Mansa
  - Hospital das Clinicas da Universidade Federal de Minas Gerais (HCUFMG), Belo Horizonte,Minas Gerais
  - SAPIENS - Instituto de Estudos e Pesquisa Clínica, Curitiba
  - CLARE - Clinica de Pneumologia, Goiânia
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Nossa Senhora da Conceição, Porto Alegre - RS
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo
- Canada (13):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Kelowna Respirology & Allergy Research, Kelowna, British Columbia
  - St. Paul's Hospital (Vancouver), Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Dr. Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Dr. Syed Anees Medicine Professional Corporation, Windsor, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - CIC Mauricie Inc., Trois-Rivières, Quebec
  - Royal University Hospital (Saskatoon), Saskatoon, Saskatchewan
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Chile (2):
  - Instituto Nacional del Tórax, Providencia, Santiago de Chile
  - Centro de Investigación del Maule, Talca
- China (37):
  - Beijing Chao-Yang Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - People's Hospital of Sichuan Province, Chengdu
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - NanFang Hosptial, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - The First hospital of Jiaxing, Jiaxing
  - Jinhua Municipal Central Hospital, Jinhua
  - Nanjing Drum Tower Hospital, Nanjing
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Huadong Hospital affiliated to Fudan University, Shanghai
  - China Shenyang Chest Hospital, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital Affiliated Tongji Medical College Huazhong University of S & T, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Second Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
  - Yichang Central People's Hospital, Yichang
  - General Hospital of Ningxia Medical University, Yinchuan
- Croatia (3):
  - University hospital center Zagreb, Zagreb
  - University Hospital Dubrava, Zagreb
  - Solmed Polyclinic, Zagreb
- University Thomayer´s Hospital, Prague, Czechia
- Denmark (2):
  - Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense C
- North Estonia Medical Centre Foundation, Tallinn, Tallinn, Estonia
- Finland (4):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - Oulun yliopistollinen keskussairaala, Oulu
  - Tampere University Hospital, Tampere
  - TYKS, Turku
- France (21):
  - HOP d'Angers, Angers
  - HOP Avicenne, Bobigny
  - HOP de la Cavale Blanche, Brest
  - HOP Louis Pradel, Bron
  - HOP CHU Caen, Caen
  - HOP François Mitterrand, Dijon
  - HOP Michallon, La Tronche
  - HOP Bicêtre, Le Kremlin-Bicêtre
  - INS Coeur Poumon, Lille
  - HOP Nord, Marseille
  - HOP Nord Laennec, Nantes
  - HOP Pasteur, Nice
  - HOP Paris Saint-Joseph, Paris
  - HOP Européen G. Pompidou, Paris
  - HOP Bichat, Paris
  - HOP Haut-Lévêque, Pessac
  - HOP Robert Debré, Reims
  - HOP Pontchaillou, Rennes
  - HOP Charles Nicolle, Rouen
  - HOP Foch, Suresnes
  - Hôpital Larrey - CHU de Toulouse, Toulouse
- Georgia (3):
  - National Center for Tuberculosis and Lung Diseases, Tbilisi, Tbilisi
  - LLC Diacor, Tbilisi
  - LTD The First Medical Center, Tbilisi
- Germany (19):
  - Velocity Clinical Research Germany GmbH, Ahrensburg, Ahrensburg
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Klinikum Region Hannover GmbH, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikum Konstanz, Konstanz
  - Klinikum der Universität München AÖR, München
  - Klinikum Nürnberg, Nuremberg
  - Krankenhaus Bethanien gGmbH, Solingen
  - Helios Hanseklinikum Stralsund, Stralsund
  - Robert Bosch Gesellschaft für medizinische Forschung mbH, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
- Greece (4):
  - Hospital of Heraklion (PAGNI), Heraklion
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - Univ. Gen. Hosp. of Patras, Pátrai
  - General Hospital of Thessaloniki "Hippokrateio", Thessaloniki
- Hungary (3):
  - Semmelweis University, Budapest
  - Koranyi National Institute For Pulmonolgy, Budapest
  - University of Debrecen Clinical Centre, Debrecen
- India (2):
  - Bhatia Hospital, Mumbai
  - P.D. Hinduja National Hospital, Mumbai
- Connolly Hospital Blanchardstown, Dublin, Ireland
- Israel (4):
  - Shamir Medical Center (Assaf Harofeh), Beer Yaakov
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Italy (13):
  - ASST degli Spedali Civili di Brescia, Brescia
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - A. O. Universitaria Careggi, Florence
  - Ospedale Colonnello D Avanzo, Foggia
  - Ospedale G.B. Morgagni, Forlì
  - Ospedale San Paolo-MILANO-18793, Milan
  - Ospedale Classificato San Giuseppe, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - A.O. San Gerardo di Monza, Monza
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - A.O.U. Senese, Siena
  - Ospedali Riuniti di Ancona, Torrette Di Ancona (Ancona)
- Japan (38):
  - Tosei General Hospital, Aichi, Seto
  - Chiba University Hospital, Chiba, Chiba
  - University of Fukui Hospital, Fukui, Yoshida-gun
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Fukuoka, Iizuka
  - Hospital of the University of Occupational and Environmental Health, Fukuoka, Kitakyushu
  - Kurume University Hospital, Fukuoka, Kurume
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Tsuboi Hospital, Fukushima, Koriyama
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Kobe City Hospital Organization Kobe City Medical Center West Hospital, Hyogo, Kobe
  - Kagawa University Hospital, Kagawa, Kita-gun
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Miyagi, Sendai
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kindai University Hospital, Osaka, Sakai
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Osaka Medical and Pharmaceutical University Hospital, Osaka, Takatsuki
  - Saitama Red Cross Hospital, Saitama, Saitama
  - Shimane University Hospital, Shimane, Izumo
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Tokushima University Hospital, Tokushima, Tokushima
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Toranomon Hospital, Tokyo, Minato-ku
  - Kyorin University Hospital, Tokyo, Mitaka
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
  - Keio University Hospital, Tokyo, Shinjuku-ku
  - National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Malaysia (4):
  - Hospital Pulau Pinang-Pulau Pinang-21953, George Town
  - Hospital Sultan Idris Shah Serdang, Kajang
  - Institut Perubatan Respiratori, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Mexico (7):
  - Centro de Investigacion Integral MEDIVEST S.C, Chihuahua City
  - CREPID Aire y Salud, Coyoacán
  - Centro de Investigacion Farmacologica del Bajío, S.C., León
  - Soltmed Smo, Mexico City
  - Centro Respiratorio de Mexico, Mexico City
  - Centro de Prevención y Rehabilitación de Enfermedades Pulmon, Monterrey
  - Oaxaca Site Management Organization, S.C., Oaxaca City
- Netherlands (4):
  - Zuyderland Medisch Centrum, HEERLENHeerlen
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam
- New Zealand (4):
  - Aotearoa Clinical Trials, Papatoetoe, Auckland
  - Waikato Hospital, Hamilton
  - Greenlane Clinical Centre, One Tree Hill, Auckland
  - Tauranga Hospital, Tauranga South
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Akershus Universitetssykehus HF, Nordbyhagen
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Poland (5):
  - University Clinical Center, Gdansk, Gdansk
  - Leszek Giec Upper-Silesian Med.Cent.Silesian Med.Univ., Katowice
  - Alergopneuma Medical Center, Świdnik
  - Nat.Instit.of Tuberculosis&LungDiseases,Outpat.Clin,warszawa, Warsaw
  - University Clinical Center of the Medical University of Warsaw, Warsaw
- Portugal (5):
  - ULS Braga, Braga
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - ULS de São José, E.P.E., Lisbon
  - USLM, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E, Vila Nova de Gaia
- King Abdullah International Medical Research Center, Riyadh, Saudi Arabia
- Serbia (3):
  - University Clinical Center of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - University Clinical Center Nis, Niš
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Hospital Golnik - Univ. Clinic of Pulmonary and Allergic Diseases, Golnik, Slovenia
- Enhancing Care Foundation NPC, Mount Edgecombe, South Africa
- South Korea (8):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (23):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital de Galdakao, Galdakao
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario De La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital General Universitario de Valencia, Valencia
- Sweden (2):
  - Universitetssjukhuset, Linköping, Linköping
  - Akademiska sjukhuset, Uppsala
- Universitätsspital Basel, Basel, Switzerland
- Taiwan (6):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - Siriraj Hospital, Bangkok Noi
  - Srinagarind Hospital, Khon Kaen
  - Maharat Nakhonchiangmai Hospital, Muang
  - Ramathibodi Hospital, Ratchatewi
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (5):
  - Gulhane Training and Research Hospital, Ankara
  - Ankara Universitesi Tip Fakultesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi -ANTALYA-33606, Antalya
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Gazi Universitesi Tip Fakultesi, Yenimahalle/ANKARA
- United Kingdom (13):
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Southmead Hospital, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Royal Lancaster Infirmary, Lancaster
  - St James's University Hospital, Leeds
  - Guy's Hospital, London
  - Royal Brompton Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Wythenshawe Hospital, Manchester
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- [Derived] Wuyts WA, Richeldi L, Assassi S, Azuma A, Cottin V, Hoffmann-Vold AM, Kreuter M, Oldham JM, Martinez FJ, Valenzuela C, Wijsenbeek MS, Kanakapura M, James A, Weimann G, Drzewuski C, Coeck C, Maher TM. Design of an open-label extension trial of nerandomilast (BI 1015550) in patients with idiopathic pulmonary fibrosis and progressive pulmonary fibrosis (FIBRONEER-ON). BMC Pulm Med. 2025 Dec 4;26(1):10. doi: 10.1186/s12890-025-03973-7. PMID 41345848
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing